CLINICAL TRIAL: NCT04115150
Title: Short-term Outcome After Ventral Hernia Repair Using Self-gripping Mesh in Subway Technique - a Retrospective Cohort Analysis
Brief Title: Short-term Outcome After Ventral Hernia Repair
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Felix Harpain, Principle Investigator, M.D., Medical University of Vienna
Other Study IDs: 1258/2018
Record Dates: First submitted 2019-10-02; First posted 2019-10-03 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Short-term Outcome After Ventral Hernia Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- self-gripping mesh
- non-self-gripping mesh

SUMMARY:
Hernia repair in sublay technique is widely accepted for ventral hernias, as it appears to be advantageous in terms of complication and recurrence rates. Recently, self-gripping meshes are increasingly used for hernia repair with retromuscular mesh positioning. However, real-life data on the safe use in that specific indication are still lacking. Therefore, this study evaluated short-term postoperative outcome of self-gripping versus conventional non-self-gripping meshes in sublay hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* ventral hernia repair in sublay technique

Exclusion Criteria:

* ventral hernia repair in other technique

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective single-centre cohort study was performed for the time period of January 2011 to July 2018. All patients, receiving a ventral hernia repair (including incisional, umbilical or epigastric hernias) in Rives-Stoppa retromuscular mesh placement technique (sublay), were included into the final analysis.
Sampling Method: Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Complication rate | 1 year
  overall complication rate, seroma rate, SSI rate

IPD SHARING:
Plan to Share IPD: No